CLINICAL TRIAL: NCT02984865
Title: The Application of Transversus Abdominis Plane Block Plus Rectus Sheath Block in Peritoneal Dialysis Catheter Placement and Analgesia Based on Transversus Abdominis Plane Block Combined With κ Receptor Agonist and NSAID(Non-steroidal Anti-inflammatory Drug ) Following Open Gastrointestinal Surgery
Brief Title: The Application of Transversus Abdominis Plane Block Plus Rectus Sheath Block in Clinical Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PJ-2016-09-05
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Nausea and Vomiting; Surgery; Anesthesia; Peritoneal Dialysis; Rectus Sheath Block
Keywords: transversus plane block; opioid; nalbuphine; gastrointestinal surgery; elderly patient; rectus sheath block; Peritoneal dialysis
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Sufentanil; Nalbuphine

STUDY DESIGN:
Intervention Model Description: The first group was designed to observe the advantage of transversus abdominis plane (TAP) block combined with rectus sheath (RS) block in PD catheter placement surgery, which is independent from other 4 groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- group S (Active Comparator): Patients were attach with PCA containing 100ml combination of sulfentanyl 2.5ug/kg and flubiprofen axetil 100mg after receiving the loading dose of sulfentanyl 5 ug and flubiprofen axetil 50mg intravenously 30 mins before the end of the operation .
  Interventions: Drug: Sulfentanyl; Drug: flubiprofen axetil
- group N1 (Experimental): Patients were attach with PCA containing 100ml combination of nalbuphine 1.5mg/kg and flubiprofen axetil 100mg after receiving the loading dose of nalbuphine 5 mg and flubiprofen axetil 50mg intravenously 30 mins before the end of the operation .
  Interventions: Drug: Nalbuphine; Drug: flubiprofen axetil
- group N2 (Experimental): Patients were attach with PCA containing 100ml combination of nalbuphine 2mg/kg and flubiprofen axetil 100mg after receiving the loading dose of nalbuphine 5 mg and flubiprofen axetil 50mg intravenously 30 mins before the end of the operation .
  Interventions: Drug: Nalbuphine; Drug: flubiprofen axetil
- group N3 (Experimental): Patients were attach with PCA containing 100ml combination of nalbuphine 2.5mg/kg and flubiprofen axetil 100mg after receiving the loading dose of nalbuphine 5 mg and flubiprofen axetil 50mg intravenously 30 mins before the end of the operation .
  Interventions: Drug: Nalbuphine; Drug: flubiprofen axetil
- Group ESRD (Other): 30 patients with ESRD who underwent PD catheter placement using left lateral transversus abdominis plane (TAP) block combined with rectus sheath (RS) block from our center. The TAP and RS blocks were respectively conducted with 15 ml of 0.5% ropivacaine and 10 ml of 0.5% ropivacaine. Pain intensity was evaluated by verbal rating scale (VRS), and the degree of patient and surgeon satisfaction was qualified by a categorical scale.
  Interventions: Procedure: rectus sheath block

INTERVENTIONS:
Drug: Sulfentanyl
  Other Names: sulfentanil
  Arms: group S
Drug: Nalbuphine
  Arms: group N1; group N2; group N3
Drug: flubiprofen axetil
  Arms: group N1; group N2; group N3; group S
Procedure: rectus sheath block — Transversus abdominis plane (TAP) block combined with rectus sheath (RS) block will be applied in Group ESRD
  Arms: Group ESRD

SUMMARY:
Peritoneal dialysis (PD) catheter placement surgery for patients with end-stage renal disease (ESRD) can be performed under peripheral nerve block. This study assessed the ability of ultrasound guided left lateral transversus abdominis plane (TAP) block combined with rectus sheath (RS) block in PD catheter placement surgery. Also, surgeries are common surgeries performed in elderly patients throughout the world. Although there is an increasing trend towards laparoscopic surgeries, open procedures continue to remain common therapeutic modalities especially in the developing countries. Pain is reported more commonly in patients undergoing open procedures than laparoscopic procedures. Postoperative pain and tissue injury associated with surgery initiated a systemic stress response which has neuroendocrine, immunological, and haematological responses. Opioids are an important modality of postoperative pain management. They blunt the neuroendocrine stress response to pain. However, they are associated with several adverse effects like respiratory depression, nausea, vomiting , pruritus, constipation, urinary retension, bradycardia and hypotension. Transversus abdominis plane block（TAPB）is a relative novel procedure in which local anesthetic agents are injected into the anatomic plane between the internal oblique and the transversus abdominis muscle. It allows a significantly prolonged duration of analgesia during the early postoperative stage in abdominal surgery. This regional anesthesia technique provides analgesia to the skin, muscles of the anterior abdominal wall and parietal peritoneum in order to decrease the incision-related pain. Thus, it reduces postoperative opiate requirements and opioids-related side effects (nausea, vomiting, delayed resumption of intestinal transit, drowsiness, respiratory depression, urine retention). Nalbuphine, being mu antagonist an kappa agonist, has a ceiling effect in its respiratory depression. Many studies have reported that incidence of adverse effects like pruritus and PONV is lower with nalbuphine in comparison with morphine. The purpose of this study is to compare the analgesic efficacy and side effect profile of sulfentanyl with nalbuphine in elderly patients undergoing open gastrointestinal surgeries.

DETAILED DESCRIPTION:
This study will be conducted in the department of Anesthesiology of the first affiliated hospital of Anhui Medical University, Hefei city, Anhui province, China. In our part 1, we are plan to observe 30 patients with ESRD who underwent PD catheter placement using left lateral transversus abdominis plane (TAP) block combined with rectus sheath (RS) block from our center. The TAP and RS blocks will be respectively conducted with 15 ml of 0.5% ropivacaine and 10 ml of 0.5% ropivacaine. Pain intensity will be evaluated by verbal rating scale (VRS), and the degree of patient and surgeon satisfaction will be qualified by a categorical scale. In part 2, the sample size was calculated based on the previous data in our hospital using sulfentanyl and flurbiprofen axetil as the opioid analgesic. The rate of postoperative nausea and vomiting(PONV) after surgery was 35%. Keeping the power of the study as 80% and 5% alpha error with the number of pairwise comparisons as 6, a total sample size of 124 was needed to identify a difference of 0.25 in the rate of PONV. Each group would require at least 31 patients. To allow for dropouts, the investigator decided to include 40 patients in each group. Elderly patients who were over 65 years old, undergoing open gastrointestinal surgeries were included in the study. Patients were divided into four groups, that is group S, group N1, group N2 and group N3, based on the drawing of an opaque sealed envelop.The anesthesiologists managing the intraoperative and postoperative courses as well as patients were blinded to the group which they belonged.The drug solution to be used intraoperatively and postoperatively as PCA (patient-controlled analgesia) was prepared by an assistant. Patients were interviewed before surgery and informed written consent was taken form each patient. Patients were shown a VAS (visual analogue score) of 0-10 for pain with 0 being no pain and 10 being worst pain ever felt, and instructed upon the use of PCA (patient-controlled analgesia) before surgery. Patients were subjected to monitoring of ECG, pulse oximetry and invasive blood pressure. 20ml combination of 0.5% ropivacaine and 10mg dexamethasone was injected bilaterally between the internal oblique and transverse abdominis muscles using sonography. All groups received standard general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD scheduled for PD catheter placement belonging to American Society of Anesthesiologists (ASA) Grade 2 to 4 were included in the study.
* Elderly patients who were over 65 years old ,undergoing open gastrointestinal surgeries were included in the study.

Exclusion Criteria:

* Exclusion criteria included patients refusal, history of abdominal surgery, coagulation disorders, allergy to local anesthetic and localized infection on the injection site.
* The exclusion criteria were patient refusal, respiratory insufficiency,cardiac insufficiency,liver or kidney dysfunction，history of brain disease,local anesthetic allergy, dysfunction of blood coagulation，hemodynamic instability, history of any chronic pain, and history of chronic opioid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2018-04-08 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 48 hours after surgery
verbal rating scale | during surgery

SECONDARY OUTCOMES:
postoperative visual analogue scale of pain | 48 hours after surgery
postoperative Ramsay of sedation | 48 hours after surgery
first time for out of bed activity after surgery | 7days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xuesheng Liu, Doctor, Study Director — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- the First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lissauer J, Mancuso K, Merritt C, Prabhakar A, Kaye AD, Urman RD. Evolution of the transversus abdominis plane block and its role in postoperative analgesia. Best Pract Res Clin Anaesthesiol. 2014 Jun;28(2):117-26. doi: 10.1016/j.bpa.2014.04.001. Epub 2014 May 9. PMID 24993433
- [Background] Zeng Z, Lu J, Shu C, Chen Y, Guo T, Wu QP, Yao SL, Yin P. A comparision of nalbuphine with morphine for analgesic effects and safety : meta-analysis of randomized controlled trials. Sci Rep. 2015 Jun 3;5:10927. doi: 10.1038/srep10927. PMID 26039709
- [Background] Kartalov A, Jankulovski N, Kuzmanovska B, Zdravkovska M, Shosholcheva M, Spirovska T, Petrusheva AP, Tolevska M, Srceva M, Durnev V, Jota G, Selmani R, Sivevski A. Effect of Adding Dexamethasone as a Ropivacaine Adjuvant in Ultrasound-Guided Transversus Abdominis Plane Block for Inguinal Hernia Repair. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2015;36(3):35-41. doi: 10.1515/prilozi-2015-0076. PMID 27442394
- [Background] Huang D, Ma X, Zhou D. [Effects of postoperative analgesia of ultrasound-guided transversus abdominis plane block in hemicolectomy patients]. Zhonghua Yi Xue Za Zhi. 2014 Jun 3;94(21):1623-6. Chinese. PMID 25152283
- [Background] Akshat S, Ramachandran R, Rewari V, Chandralekha, Trikha A, Sinha R. Morphine versus Nalbuphine for Open Gynaecological Surgery: A Randomized Controlled Double Blinded Trial. Pain Res Treat. 2014;2014:727952. doi: 10.1155/2014/727952. Epub 2014 Apr 14. PMID 24834352
- [Derived] Dai W, Lu Y, Liu J, Tang L, Mei B, Liu X. Ultrasound-guided left lateral transversus abdominis plane block combined with rectus sheath block in peritoneal dialysis catheter placement. J Anesth. 2018 Aug;32(4):645-648. doi: 10.1007/s00540-018-2528-2. Epub 2018 Jul 5. PMID 29978298
- [Derived] Mao Y, Cao Y, Mei B, Chen L, Liu X, Zhang Z, Gu E. Efficacy of Nalbuphine with Flurbiprofen on Multimodal Analgesia with Transverse Abdominis Plane Block in Elderly Patients Undergoing Open Gastrointestinal Surgery: A Randomized, Controlled, Double-Blinded Trial. Pain Res Manag. 2018 Jan 28;2018:3637013. doi: 10.1155/2018/3637013. eCollection 2018. PMID 29623143